CLINICAL TRIAL: NCT04252261
Title: Effects of Sulforaphane on Cognitive Function in Patients With Frontal Brain Damage: Study Protocol for a Randomized Controlled Trial
Brief Title: Effects of Sulforaphane on Cognitive Function in Patients With Frontal Brain Damage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202001005
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Frontal Lobe Dysfunction
Keywords: Sulforaphane; frontal brain damage; cognitive deficits; cognitive function; brain metabolites; gut microbiota
MeSH Terms: conditions — Cognition Disorders | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and researchers are blind to the treatment allocation (double-blind). An independent researcher developed the computer-generated randomization plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sulforaphane (Experimental): To evaluate the effect of sulforaphane treatment on the cognitive deficits of patients with frontal brain damage
  Interventions: Drug: sulforaphane
- placebo (Placebo Comparator): To evaluate the effect of sulforaphane treatment on the cognitive deficits of patients with frontal brain damage
  Interventions: Drug: placedo

INTERVENTIONS:
Drug: sulforaphane — To evaluate the effects of sulforaphane on the cognitive improvement of patients with frontal brain damage
  Arms: sulforaphane
Drug: placedo — To evaluate the effects of sulforaphane on the cognitive improvement of patients with frontal brain damage
  Arms: placebo

SUMMARY:
High rates of patients with frontal brain damage show serious cognitive functional deficits, which negatively impact their quality of life and are linked with poor clinical outcomes. Sulforaphane has shown significant antioxidant and cellular protective effects in animal models associated with oxidative stress, such as focal cerebral ischemia, brain inflammation, and intracranial hemorrhage. Preclinical research has shown that sulforaphane can significantly improve spatial localization and working memory impairment after brain damage. The primary aim of this clinical trial is to assess the efficacy of sulforaphane for improving cognitive function in patients with frontal brain damage.

DETAILED DESCRIPTION:
90 patients aged 18-65 years, of both genders, who have incurred cognitive deficits after frontal brain damage will be recruited in the neurosurgery department in Xiangya hospital. All focal lesions were confined to the frontal brain, which is verified by CT or MRI. Cognitive deficits will be diagnosed using the Chinese version of the Montreal Cognitive Assessment (MoCA-C). All eligible recruited patients will be randomly divided into two groups in a 2:1 ratio. Participants will receive a battery of cognitive tests at baseline and again after 4 and 12 weeks to determine the effect of sulforaphane on cognition. T1-weighted brain magnetic resonance images and resting-state functional MRI will be carried out using 3 Tesla (3T) brain MRI at these timepoints. Brain magnetic resonance spectrum will be applied to detect MRI markers of brain metabolites and gut microbiota will also be assessed over this period.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Focal lesions were confined to the frontal brain, which is verified by CT or MRI
* Clinical diagnosis of Cognitive deficits using the Chinese version of the Montreal Cognitive Assessment (MoCA-C) with scores < 26 will be assessed as having cognitive deficits (<25 for patients educated <12 years)
* be adherent to the continued sulforaphane treatment medication

Exclusion Criteria:

* Previous history of cognitive impairment
* Brain MRI indicating damage was not restricted to the frontal lobe.
* Inability to cooperate with cognitive testing for disturbance of consciousness or mental disorder
* Pregnancy or maternal lactation
* Life expectancy < 3 months
* CO poisoning, autoimmune encephalitis, intracranial infection, or other types of diffuse intracranial disease.
* plan to receive radiotherapy during the trial period
* Laboratory examination showing liver and kidney insufficiency or other severe complications; the presence of diseases which may interfere with the results of the evaluation
* Involvement in other trials 1 month prior to the start of the trial or during the trial period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline cognitive tests scores at 3 months | Week 1 and week 12.
  The battery of cognitive tests include different domains of cognitive tests, higher scores indicates better cognition.

SECONDARY OUTCOMES:
the resting state MRI (rsMRI) | Week 0 and 12.
  It can be served as a powerful tool to map networks of "functional connectivity" in the brain even in the absence of task activation or stimulation.
T1-weighted spin-echo MRI | Week 0, 4, and 12.
  It can be used as outcome measures in therapeutic trials

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and informed consent form are available on request to the corresponding author.
Supporting Information: Study Protocol, ICF
Time Frame: 2021-2022
Access Criteria: The sharing data for this study are available on request to the corresponding author

REFERENCES:
- [Derived] Liu F, Huang J, Hei G, Wu R, Liu Z. Effects of sulforaphane on cognitive function in patients with frontal brain damage: study protocol for a randomised controlled trial. BMJ Open. 2020 Oct 16;10(10):e037543. doi: 10.1136/bmjopen-2020-037543. PMID 33067279